CLINICAL TRIAL: NCT05881824
Title: PAP Treatment Adherence Supported by Dietary Intervention Isimproved in Overweight and Obese Obstructive Sleep Apnea(OSA) Patients: A Randomized, Controlled Trial
Brief Title: PAP Adherence After Diet/Lifestyle Intervention in OSA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Izolde Bouloukaki, Clinical Researcher, University of Crete
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSADIET1
Record Dates: First submitted 2023-05-19; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; treatment adherence; Positive airway pressure (PAP) treatment; diet/lifestyle intervention; Mediterranean diet
MeSH Terms: conditions — Sleep Apnea, Obstructive; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care group (SCG) (No Intervention): The SCG received oral healthy lifestyle advice and counseling on physical activity and sleep habits
- Mediterranean diet group (MDG) (Active Comparator): The MDG was additionally subjected to a 6-month behavioral intervention aiming at weight loss and increasing adherence to the Mediterranean diet.
  Interventions: Behavioral: MDG intervention

INTERVENTIONS:
Behavioral: MDG intervention — 6-month behavioral intervention aiming at weight loss and increasing adherence to the Mediterranean diet
  Arms: Mediterranean diet group (MDG)

SUMMARY:
The aim of this study is to explore the role of diet/lifestyle intervention on Positive airway pressure (PAP) treatment adherence in patients with obstructive sleep apnea (OSA).Specifically, we evaluated the effects of a combination of PAP and weight-loss Mediterranean diet intervention on improving PAP adherence, Body mass index (ΒΜΙ), daytime symptoms, mainly sleepiness and arterial blood pressure measurements over the effect of standard care alone.

DETAILED DESCRIPTION:
We designed a parallel, randomized, controlled, clinical trial. Eligible participants are adult, overweight and obese men and women, diagnosed with moderate-to-severe OSA [apnea-hypopnea index (AHI)≥15 events/h] through an attended overnight polysomnography. Participants, after written informed consent, were blindly randomized to a standard care group (SCG, n=37) and a Mediterranean diet group (MDG, n=37). Study groups were prescribed PAP. The SCG received oral healthy lifestyle advice and counseling on physical activity and sleep habits, while the MDG was additionally subjected to a 6-month behavioral intervention aiming at weight loss and increasing adherence to the Mediterranean diet. PAP adherence (hours of device use), BMI, daytime sleepiness, evaluated by Epworth Sleepiness Scale (ESS) and arterial blood pressure measurements were evaluated pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with newly diagnosed moderate to severe OSA [apnea-hypopnea index (AHI)≥15 events/h] through an attended overnight polysomnographyaccording to standard criteria
* overweight and obese [BMI>25 kg/m2]
* eligible for PAP treatment with adherence data available in the 6-months after initiation of treatment and
* with an above-elementary school education.

Exclusion Criteria:

* refusal to participate
* patients on PAP treatment
* current participation in a weight loss program
* central sleep apnea syndromes
* obesity hypoventilation syndrome
* restrictive ventilator syndromes
* severe congestive heart failure
* a history of life-threatening arrhythmias
* severe cardiomyopathy
* long-term oxygen therapy
* chronic kidney disease
* family or personal history of mental illness
* drug or alcohol abuse
* severe cognitive impairment
* concurrent oncological diseases
* pregnancy or lactatio
* recent hospitalization for acute or chronic respiratory disease
* history of narcolepsy or restless leg syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Difference in PAP adherence | 6 months
  Difference pre post in PAP adherence (hours of device use)

SECONDARY OUTCOMES:
Difference in Body mass index | 6 months
  Difference pre post intervention in Body mass index
Difference in Blood pressure measurements | 6 months
  Difference in Systolic and Diastolic Blood pressure measurements pre and post intervention
Difference in daytime sleepiness | 6 months
  Difference ipre post intervention in daytime sleepiness assessed by Epworth Sleepiness Scale score

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Schiza, MD, Study Chair — University of Crete
Locations (1):
- University of Crete, Heraklion, Crete, Greece

IPD SHARING:
Plan to Share IPD: No